CLINICAL TRIAL: NCT01492556
Title: A Phase II, Single-arm, Multicenter Study of Etoposide Monotherapy in Treating Patients With Recurrent or Metastatic Breast Cancer
Brief Title: Study of Etoposide in Treating Patients With Recurrent or Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Peking Union Medical College Hospital (Other); Beijing Chao Yang Hospital (Other); China-Japan Friendship Hospital (Other); Beijing Hospital of the Ministry of Health (Unknown); The First Affiliated Hospital of Dalian Medical University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Zhejiang Cancer Hospital (Other); Henan Cancer Hospital (Other Government); Guangxi Cancer Hospital (Unknown); Shanghai Putuo District Center Hospital (Other); International Peace Maternity and Child Health Hospital (Other); Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Binghe Xu, Deputy Director of Department of Medical Oncology, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-BC-015
Record Dates: First submitted 2011-12-12; First posted 2011-12-15 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer
Keywords: Recurrent; Metastatic; Breast cancer
MeSH Terms: conditions — Breast Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etoposide (Experimental): Etoposide Capsules
  Interventions: Drug: Etoposide

INTERVENTIONS:
Drug: Etoposide — Lastet (Etoposide Capsules, 25mg*40 capsules/box), manufactured by Nippon Kayaku Co., Ltd.
  Other Names: Lastet, VP-16

SUMMARY:
The purpose of this study is to determine whether Etoposide Monotherapy is effective and safe in the treatment of recurrent or metastatic breast cancer in Chinese female patients.

DETAILED DESCRIPTION:
Current recommended dosage of Etoposide in treating breast cancer is 50 mg/m2 orally once a day for 21 days, repeated every 28 days. With retrospective data review, this study intends to adjust Etoposide dose to 60 mg/m2 daily for 10 days, repeated every 21 days as a cycle, to investigate the effectiveness and safety of Etoposide monotherapy in the treatment of recurrent or metastatic breast cancer in Chinese female patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years old.
* ECOG status: 0-2.
* Histologic or cytologic diagnosis of locally advanced or metastatic breast cancer.
* No more than three prior chemotherapies, adjuvant chemotherapy excluded.
* Received prior anthracycline, taxane therapy.
* At least 4 weeks from previous chemotherapy.
* Measurable disease of >=2 cm (>=1 cm on spiral CT scan).
* Life expectancy of ≥ 3 months.
* Adequate organ functions:

  * Hemoglobin ≥10.0 g/dl, Absolute neutrophil count ≥1.5×10^9/L, Platelet count ≥100×10^9/L,
  * Creatinine clearance ≥60ml/min,
  * Bilirubin ≤1.5 times upper limit of normal (ULN); AKP,AST and ALT ≤2.5x ULN(≤5x ULN if due to liver metastases).
* Signed informed consent.
* Menopausal women or received surgical sterilization, women with children potential must not be pregnant or nursing with negative pregnancy test and willing to practice acceptable methods of birth control during the study and 3 months after the study.

Exclusion Criteria:

* Pregnancy or lactation.
* Untreated or uncontrolled CNS metastases, or with refractory psychiatric illness.
* Prior treatment with Etoposide.
* Other primary malignancies within the past 5 years except for carcinoma in situ of the cervix or nonmelanoma skin cancer.
* Clinically significant heart diseases (e.g.congestive heart failure, symptomatic coronary disease, uncontrolled cardiac arrhythmia, Myocardial infarction) within the past 12 months.
* Serious uncontrolled concurrent infection or metabolism disorder.
* Concurrent treatment for active peptic ulcer disease or with digestive disorders.
* Prior radiotherapy and major surgery within 3 weeks before screening.
* Less than 4 weeks since prior investigational agents.
* Metastases present in more than one-third whole liver.
* Unable or unwilling to comply with the study protocol.
* Unsuitable to participate in study, that in the opinion of the treating physician.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Up to 1 year

SECONDARY OUTCOMES:
Clinical response rate | Every six weeks
  Assessed by RECIST v1.1 criteria.
1-year survival rate | Up to 1 year
Adverse events | Subjects will be followed from date of enrollment until the date of last visit, expected up to 1 year
Quality of Life | Every six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, M.D., Ph.D, Principal Investigator — Chinese Academy of Medical Sciences
Locations (14):
- China (14):
  - Beijing Hospital of the Ministry of Health, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Chao-yang Hospital, Beijing, Beijing Municipality
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Guangxi Cancer Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - International Peace Maternity & Child Health Hospital of the China Welfare Institute, Shanghai, Shanghai Municipality
  - Shanghai Putuo District Center Hospital, Shanghai, Shanghai Municipality
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang